CLINICAL TRIAL: NCT00067249
Title: Women's Use of Alternative Medicine: A Multiethnic Study
Status: Completed | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Other Study IDs: F31AT001401-01 (NIH)
Record Dates: First submitted 2003-08-13; First posted 2003-08-15 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2007-02

CONDITIONS: Uterine Fibroids; Osteoporosis; Urinary Tract Infection; High Blood Pressure; Heart Disease; Arthritis; Depression; Headaches
Keywords: Race; Ethnicity; Complementary and Alternative Medicine; Women's health; Social determinants of Health
MeSH Terms: conditions — Leiomyoma; Osteoporosis; Urinary Tract Infections; Hypertension; Heart Diseases; Arthritis; Depression; Headache

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
The purpose of this study is to examine socio-cultural factors of women's use of complementary and alternative medicine (CAM). The effects of socioeconomic status, social networks and acculturation on CAM use will be assessed among white, African-, Mexican-, and Chinese-American women.

ELIGIBILITY:
Inclusion criteria:

Experienced one or more of the following health conditions within the last year:

* pregnancy related symptoms
* menopausal related symptoms
* headaches
* back pain
* osteoporosis
* cancer
* high blood pressure
* high cholesterol
* heart disease
* joint pain/arthritis
* insomnia
* uterine fibroids
* urinary tract infection
* vaginal tract infection
* medically diagnosed depression
* menstrual symptoms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3200
Dates: Start 2001-04; Study Completion 2001-09

CONTACTS AND LOCATIONS:
Overall Officials: Fredi Kronenberg, PhD, Principal Investigator — Rosenthal Center for Complementary and Alternative Medicine, Columbia University